CLINICAL TRIAL: NCT04657120
Title: Safety and Efficiency of the YEARS Algorithm Versus Computed Tomography Pulmonary Angiography Alone for Suspected Pulmonary Embolism in Patients With Malignancy : HYDRA Study
Brief Title: Safety and Efficiency of the YEARS Algorithm Versus Computed Tomography Pulmonary Angiography Alone for Suspected Pulmonary Embolism in Patients With Malignancy
Acronym: HYDRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Antwerp (Other); University Hospital, Geneva (Other); Reinier de Graaf Groep (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Diakonessenhuis, Utrecht (Other); Amphia Hospital (Other); Centre Hospitalier Universitaire Vaudois (Other); Hospital Universitario Ramon y Cajal (Other); Tergooi Hospital (Other); Radboud University Medical Center (Other); Bernhoven Hospital (Other); Hôpital Louis Mourier (Other); Medisch Spectrum Twente (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Maasstad Hospital (Other); Flevo Ziekenhuis, Almere (Unknown); Groene Hart Ziekenhuis (Other); University Hospital, Brest (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Erik Klok, pr, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYDRA (NL68754.058.19)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Embolism; Embolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases; Cancer; Diagnosis
MeSH Terms: conditions — Pulmonary Embolism; Embolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases; Neoplasms; Disease | interventions — 4-((1,4,8,11-tetraazacyclotetradec-1-yl)methyl)benzoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YEARS algorithm (Experimental): Patients randomized to this arm will be evaluated according to the YEARS algorithm.
  Interventions: Procedure: YEARS algorithm
- CTPA as single test (Active Comparator): Patients randomized to this arm will undergo a contrast enhanced CTPA.
  Interventions: Procedure: CTPA

INTERVENTIONS:
Procedure: YEARS algorithm — Patients randomized to the YEARS algorithm will be evaluated according to the YEARS algorithm consisting of three items of the original Wells rule (clinical signs of DVT, haemoptysis and 'PE most likely diagnosis') and a D-dimer test. In patients without any of the three items and a D-dimer level <1.0 μg/mL (<1000ng/mL), and in patients with ≥1 items and a D-dimer level <0.5 μg/mL (<500 ng/mL) a PE is excluded without CTPA. In the other patients a standard contrast enhanced CTPA will be performed according to local practice. PE is defined as at least one filling defect in the pulmonary artery tree on CTPA.
  Arms: YEARS algorithm
Procedure: CTPA — Patients randomized to the CTPA management group will undergo a contrast enhanced CTPA to rule out PE according to standard local practice.
  Arms: CTPA as single test

SUMMARY:
The aim of this study is to prospectively validate the safety and efficiency of management according to the YEARS algorithm to safely rule out clinically suspected PE in patients with active malignancy to be compared with 'standard' management by computed tomography pulmonary angiography (CTPA) alone in a randomized study.

DETAILED DESCRIPTION:
Recently, the YEARS-algorithm was demonstrated to be a safe and efficient diagnostic strategy for patients with clinically suspected pulmonary embolism (PE). It is recognized that diagnostic algorithms for pulmonary embolism (PE) may not be as effective and safe in patients with malignancy, due to the low specificity of D-dimer test in that setting. A diagnostic algorithm that could safely rule out PE in patients with malignancy without performing computed tomography pulmonary angiography (CTPA) could nonetheless improve patient care.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Clinically suspected PE as judged by the treating clinician
* Any type of active malignancy (other than basal-cell or squamous-cell carcinoma of the skin), defined as diagnosis within six months before the study inclusion (as confirmed histologically or high suspicion as judged by the clinician), receiving treatment for malignancy at time of inclusion or during 6 months prior to randomization, including recurrent or local metastatic malignancy
* Outpatients and hospitalized patients
* Age ≥ 18 years
* Signed and dated informed consent, available for start of the trial procedure

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Medical or psychological condition that would not permit completion of the study or signing of informed consent, including life expectancy less than 3 months, or unwillingness to sign informed consent
* Treatment with full-dose therapeutically dosed anticoagulation that was initiated 24 hours or more prior to eligibility assessment
* Contraindication to CTPA

  * contrast allergy

Hemodynamic instability at presentation (as a consequence of concurrent acute PE or otherwise), indicated by at least one of the following:

* systolic blood pressure (SBP) < 100 mm Hg, or heart rate >120 beats per minute or SBP drop by > 40 mm Hg, for > 15 min
* need for catecholamines to maintain adequate organ perfusion and a systolic blood pressure of > 100 mmHg
* Need for cardiopulmonary resuscitation
* Inability to follow-up
* Life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-08-23 (Actual); Study Completion 2025-08-23 (Actual)

PRIMARY OUTCOMES:
Recurrent PE | 3 months
  Recurrent PE will be observed
Deep vein thrombosis (DVT) | 3 months
  Number of DVT will be observed
Mortality | 3 months
  The mortality will be observed Adjudicated according to ISTH definition in which both PE-related death as well as unexplained death will count towards primary outcome

SECONDARY OUTCOMES:
CTPA | 3 months
  Number of performed CTPA will be observed in the YEARS-group at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Menno Huisman, Pr, Principal Investigator — Leiden University Medical Center
Locations (28):
- Belgium (3):
  - Antwerpen University Hospital (UZA), Antwerp
  - Cliniques Universitaires Saint-Luc (CUSL), Brussels
  - Centre Hospitalier Universitaire de Liège (CHU Liège), Liège
- France (5):
  - CHU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Louis Mourier - APHP, Colombes
  - HEGP, Paris
  - CHU Saint-Etienne, Saint-Etienne
- Italy (2):
  - Policlinico di Milano Ospedale Maggiore | Fondazione IRCCS Ca' Granda, Milan
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Netherlands (14):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Flevoziekenhuis, Almere Stad
  - Amsterdam UMC, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Groene Hart Ziekenhuis, Gouda
  - Tergooi MC, Hilversum
  - Leiden University Medical Center, Leiden
  - Radboud UMC, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - Bernhoven Ziekenhuis, Uden
  - Diakonessenhuis, Utrecht
- Hospital Universitario Ramón y Cajal, Madrid, Spain
- Switzerland (3):
  - The Inselspital Bern, Bern
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by an internal committee . Requestors will be required to sign and complete a data access agreement.